CLINICAL TRIAL: NCT07052682
Title: A Multicenter, Single-arm, Open-label, Phase 1b Study to Explore the Mechanism of Action and Evaluate the Safety of Ontamalimab in Participants With Nonalcoholic Steatohepatitis With Fibrosis Stage 1 Through 4
Brief Title: A Study to Evaluate How Ontamalimab Works and Assess Its Safety and Tolerability in People With Nonalcoholic Steatohepatitis With Fibrosis Stages 1 to 4
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was terminated early by the sponsor due to a strategic shift and reprioritization of clinical programs within Takeda.
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAK-647-1001
Record Dates: First submitted 2025-06-30; First posted 2025-07-06 (Actual); Results first posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Steatohepatitis
Keywords: Drug Therapy
MeSH Terms: conditions — Fatty Liver | interventions — ontamalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ontamalimab (Experimental): Participants receive ontamalimab 75 milligrams (mg) subcutaneous (SC) injection using a prefilled syringe once every 4 weeks (Q4W) on Day 1 and the last dose is administered at Week 20 with a total treatment period of 24 weeks.
  Interventions: Drug: Ontamalimab

INTERVENTIONS:
Drug: Ontamalimab — Ontamalimab SC injection.
  Other Names: SHP647; PF-00547659; TAK-647

SUMMARY:
The main aim of this study is to evaluate the safety and tolerability of ontamalimab in participants with a liver disease called nonalcoholic steatohepatitis (NASH) or metabolic dysfunction-associated steatohepatitis (MASH) with scarring in the liver (fibrosis stage 1 to 4). The study will also check if there are any important changes in the body's health markers (biomarkers) from the beginning of the study to see if ontamalimab stops liver scarring and reduces inflammation of the liver.

Participants will be in the study for approximately up to 46 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. The participant is willing and able to understand and fully comply with study procedures and requirements, in the opinion of the investigator.
2. The participant and/or the participant's legally acceptable representative has provided informed consent (that is, in writing, documented via a signed and dated informed consent form [ICF] or electronic consent [eConsent] if applicable) and any required privacy authorization prior to the initiation of any study procedures.
3. The participant is aged 18 to 70 years, inclusive, at the time of signing the ICF.
4. The participant has signs of fibrogenic activity (Pro-C3 greater than or equal to [>=] 12.6 nanograms per milliliter [ng/mL], ELF score >=7.7) at the Week -8 (screening visit 1 [SV1]) (applies to all participants regardless of whether historical biopsy results are available at screening).
5. The participant has indication of NASH via biopsy (Nonalcoholic fatty liver disease activity score [NAS] >=3 with at least 1 point in lobular inflammation) and liver fibrosis stage 1 (F1) through fibrosis stage 4 compensated cirrhotic (F4cc) according to NASH Clinical Research Network (CRN).
6. The participant is a male participant or a nonpregnant, nonlactating female participant who, if sexually active, agrees to comply with the contraceptive requirements of the protocol, or a female participant of nonchildbearing potential. Participants of reproductive potential who are sexually active must agree to use appropriate contraception (that is, highly effective methods for female participants and medically appropriate methods for male participants) for the duration of the study and for at least 12 weeks after the last dose of study drug.
7. The participant, if capable of breastfeeding, agrees to forego breastfeeding for the period from informed consent until 12 weeks after the last dose of study drug.

Exclusion Criteria:

1. The following laboratory findings are exclusionary for all participants if found during screening visits (Week -8 [SV1], Week -6 [SV2] or at Day -4 visit [Visit 4a2]):

   1. Aspartate aminotransferase (AST) levels greater than (>) 5*the upper limit of normal (ULN).
   2. Alanine aminotransferase (ALT) levels >5*ULN.
2. The following laboratory findings are exclusionary for all participants if found during either screening visit (SV1 or SV2):

   1. Alkaline phosphatase (ALP) >=2*ULN.
   2. Serum creatinine >=1.5*ULN or has an estimated glomerular filtration rate (eGFR) less than (<) 45 milliliters per minute per 1.73 square meters (mL/min/1.73 m^2).
   3. International normalized ratio (INR) >=1.3 (except for participants who are receiving anticoagulant treatment).
   4. Total bilirubin level (TBL) >=ULN (except for participants with a documented history of Gilbert's syndrome if direct bilirubin is within normal reference range).
   5. Direct bilirubin >=3*ULN.
   6. Platelet count <60*10^9 per liter (/L).
3. The participant has been diagnosed with decompensated liver disease, or has new signs of decompensation and/or clinically meaningful change in disease status based on the judgment of the investigator (including but not limited to clinically significant changes in TBL, albumin, INR, creatinine, and/or AST and ALT levels) are observed during the screening period, or has any of the following during screening period:

   1. Presence or history of ascites, hepatic encephalopathy, or variceal bleeding.
   2. Presence or history of Child-Pugh >6 (Class B or C), unless due to therapeutic anticoagulation.
   3. Presence or history of model for end-stage liver disease (MELD) score >12. Note: It is the investigator's decision, in consultation with the sponsor, to allow participants to enter the study who have clinically meaningful rising tendencies in liver chemistries or significantly elevated liver chemistries that do not yet satisfy Exclusion Criterion #1 but could be interpreted as clinically concerning (that is, AST or ALT >4*ULN) at any visit during the screening period.
4. The participant has other diagnosed causes of liver disease based on medical history and/or baseline evaluation of laboratory and/or histology results, including, but not limited to viral (example, chronic hepatitis B, hepatitis B virus surface antigen [HBsAg] positive, or hepatitis B core antibody [HBcAB] positive; or chronic hepatitis C or hepatitis C virus antibody [HCVAb] positive and hepatitis C [HCV] ribonucleic acid [RNA] positive; or human immunodeficiency virus [HIV]-antibody positive), alcoholic (alcohol consumption greater than 4 units on any day or 14 units per week for male participants, or greater than 3 units on any day or 7 units per week for female participants [1 unit of alcohol is present in one 12 ounces [oz]/355 milliliters [mL] beer (approximately 5 percentage [%] alcohol), one 5 oz/148 mL glass of wine (approximately 12% alcohol), and one 1.5 oz/44 mL measure of 80-proof liquor (approximately 40% alcohol)]), or autoimmune conditions (example, primary sclerosing cholangitis, primary biliary cirrhosis, autoimmune hepatitis, drug-induced hepatotoxicity), and other rare liver disease (example, alpha-1-antitrypsin deficiency, Wilson disease, hemochromatosis). Note: If a participant tests negative for HBsAg but positive for HBcAb, the participant would be considered eligible if no presence of hepatitis B virus (HBV) deoxyribonucleic acid (DNA) is confirmed by HBV DNA polymerase chain reaction (PCR) reflex testing performed by the central laboratory. Participants who are HCVAb positive without evidence of HCV RNA may be considered eligible (spontaneous viral clearance or previously treated and cured [defined as no evidence of HCV RNA at least 12 weeks before baseline]).
5. The participant has a history of impaired hemostasis that, in the investigator's judgement, would increase the risk to the participant if he or she participates in the study.
6. The participant has a significant concurrent medical condition at the time of screening or baseline, including, but not limited to, the following:

   1. Any major illness/condition or evidence of an unstable clinical condition (example, hepatic, renal, hematologic, gastrointestinal, endocrine [example, uncontrolled diabetes or type 1 diabetes mellitus, or thyroid disease], neurological [pre-existing demyelinating disorder such as multiple sclerosis or new onset seizures, unexplained sensory motor, or cognitive behavioral, neurological deficits, or significant abnormalities noted during screening], cardiovascular, pulmonary, immunologic [example, Felty's syndrome], or local active infection/infectious illness [any bacterial, fungal, or viral, example, clinically active cytomegalovirus, Epstein-Barr virus, herpes simplex virus]) that, in the investigator's judgment will substantially increase the risk to the participant if he or she participates in the study.

      Note: Participants with hemoglobin A1c (HbA1c) of >=6.5% at screening (SV1; Week -8) without a previous diagnosis of type 2 diabetes mellitus (T2DM) should be excluded from the study. Participants with a previous diagnosis for T2DM are permitted to enter the study if on a stable regimen of antidiabetic therapy for at least 90 days before screening. Participants who are on a stable regimen of antidiabetic therapy for at least 90 days before screening (SV1; Week -8) and have HbA1c of >=9% at Week -8 (SV1) should be excluded.
   2. Presence of acute coronary syndrome (example, acute myocardial infarction, unstable angina pectoris) within 24 weeks before screening.
   3. History of significant cerebrovascular disease within 24 weeks before screening.
   4. Cancer or history of cancer, including hepatocellular carcinoma or cholangiocarcinoma, or lymphoproliferative disease within the previous 5 years (other than resected cutaneous basal cell carcinoma, squamous cell carcinoma, or carcinoma in situ of the uterine cervix that has been treated with no evidence of recurrence).
   5. Any other severe acute or chronic medical or psychiatric condition or laboratory or ECG abnormality that may increase the risk associated with study participation or study drug administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this study.
   6. Transplanted organ or history of liver transplantation.
   7. Significant trauma or major surgery within 4 weeks before the first screening visit, or with any major elective surgery planned to occur during the study.
7. The participant has severe active inflammatory bowel disease (IBD). Participants with inactive IBD or active of mild to moderate severity that was documented either by prior endoscopy or in previous medical records for >6 months are permitted to enter if they do not require biological treatment or Janus kinase (JAK) inhibitors. Treatment with leukocyte apheresis or selective lymphocyte, monocyte, or granulocyte apheresis or plasma exchange 30 days before baseline (Day 1).
8. The participant has a severe immune-mediated inflammatory disease (IMID) (example, rheumatoid arthritis, spondylarthritis disease spectrum, connective tissue disorders, cutaneous inflammatory conditions such as psoriasis, atopic dermatitis, hidradenitis suppurativa, asthma, multiple sclerosis). Participants with inactive IMID or active IMID of mild to moderate severity are permitted to enter the study.
9. The participant has a change in body weight >=5% three months before start of the screening or after qualifying liver biopsy. If the participant had a liver biopsy within 24 weeks of screening but experienced a weight change of >=5% since the date of liver biopsy, the liver biopsy must be repeated at screening.
10. The participant has any laboratory abnormality or condition that, in the investigator's opinion, could adversely affect the safety of the participant or impair the assessment of study results.
11. The participant has known hypersensitivity to ontamalimab or formulation excipient.
12. The participant has active or latent infection with mycobacterium tuberculosis (TB) who have not completed a generally accepted full course of treatment before screening.
13. The participant has clinically significant abnormal chest X-ray findings at SV1 (or up to 12 weeks before the first screening visit if available), such as presence of active TB, general infections, heart failure, or malignancy.
14. The participant has a positive interferon-gamma release assay (IGRA) at screening or within 12 weeks before screening even in the absence of previously diagnosed active or latent TB. IGRA screening may be repeated during the screening period if the initial result is indeterminate. The participant may be enrolled if confirmatory IGRA results from the central laboratory are negative. If the confirmatory IGRA results from the central laboratory are positive, the participant should be screen-failed. If both initial and confirmatory IGRA results are indeterminate, the participant may be enrolled after a Mantoux tuberculin skin test is negative and after consultation with the sponsor and a pulmonary or infectious disease specialist who determines low risk of infection (example, the participant would be acceptable for immunosuppressant [example, anti-tumor necrosis factor (TNF) treatment] without additional action). If the time for consultation exceeds the visit window, the participant should be screen-failed and can be rescreened after the consultation establishes eligibility for study participation. This consultation must be included in the participant's medical history.
15. The participant has any unexplained symptoms suggestive of progressive multifocal leukoencephalopathy (PML) based on the targeted neurological assessment during the screening period.
16. The participant has HIV.
17. The participant has a medical condition (example, morbid obesity, claustrophobia) that prevent execution of protocol procedures including percutaneous liver biopsy, liver stiffness measurement (LSM) by FibroScan, and magnetic resonance imaging (MRI).
18. The participant is receiving treatment with vitamin E, thiazolidinediones, or glucagon-like peptide-1 receptor agonists (GLP-1 RA) unless on a stable dose for 3 months before qualifying liver biopsy and not initiated after qualifying liver biopsy and is anticipated to maintain the same dosing regimen throughout study participation.
19. The participant is using drugs, herbs, or supplements historically associated with causing or worsening nonalcoholic fatty liver disease (NAFLD)/NASH within 24 weeks before qualifying liver biopsy or any time after qualifying liver biopsy is performed, including the use of total parenteral nutrition.
20. The participant has a positive urine screen for amphetamines, cocaine, or opioids related to the use of these drugs at screening.
21. The participant is receiving methadone or buprenorphine unless on stable maintenance treatment for at least 6 months before screening. Participants with a positive urine drug screen due to prescription opioid-based medication are eligible if the prescription and diagnosis are reviewed and approved by the investigator.
22. The participant is using any prohibited concomitant medications as described in the protocol.
23. The participant has received a live (attenuated) vaccine within 4 weeks before baseline or is anticipated to receive a live vaccine during the study.
24. The participant has participated in another investigational study of a drug or device within 30 days before or within 5 half-lives of the prior investigational agent (whichever is longer) before baseline (Day 1).
25. The participant has participated in another investigational study targeting NASH, type 2 diabetes mellitus, or obesity within 6 months before baseline (Day 1).
26. The participant is concurrently participating in another therapeutic clinical study.
27. The participant has previously received ontamalimab.
28. The participant has had previous exposure to anti-integrin or anti-adhesion molecule treatment example, natalizumab, efalizumab, etrolizumab, vedolizumab, or any other investigational anti-integrin/adhesion molecule within 90 days before baseline (Day 1).
29. The participant has had previous exposure to any other biologic drugs with immunomodulatory properties such as anti-TNF, including biosimilars or anti-interleukin (IL)-12/23, or any nonbiologic treatment with immunomodulatory properties such as JAK inhibitors within 90 days or 5 half-lives (whichever is longer) before baseline (Day 1).
30. The participant is unavailable for follow-up assessment or investigator concern for participant's compliance with the protocol procedures.
31. The participant is a study site employee, an immediate family member (example, spouse, parent, child, sibling), or is in a dependent relationship with a study site employee who is involved in conduct of this study or may consent under duress.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2023-01-18 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (15):
- United States (15):
  - Arizona Liver Health, Chandler, Arizona
  - Adobe Clinical Research, LLC, Tucson, Arizona
  - Southern California Research Center, Coronado, California
  - University of California, San Diego, NAFLD Research Center, La Jolla, California
  - California Liver Research Institute, Pasadena, California
  - Inland Empire Clinical Trials, LLC, Rialto, California
  - Covenant Metabolic Specialist LLC, Fort Myers, Florida
  - Covenant Metabolic Specialist LLC, Sarasota, Florida
  - Tandem Clinical Research GI, LLC, Marrero, Louisiana
  - Lucas Research, Inc, Morehead City, North Carolina
  - The Liver Institute at Methodist Dallas Medical Center, Dallas, Texas
  - Houston Research Institute, Houston, Texas
  - Texas Liver Institute, San Antonio, Texas
  - Pinnacle Clinical Research LLC, San Antonio, Texas
  - VCU Dept of Internal Medicine, Division of GI, Hepatology & Nutrition, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data from this particular study will not be shared as there is a reasonable likelihood that individual patients could be re-identified (due to the limited number of study participants/study sites, …)

REFERENCES:
- See also: Click here for more information about this trial in easy-to-understand language, including a Plain Language Summary of the results if the trial has been completed. — https://clinicaltrials.takeda.com/study-detail/b21025249c9a4086??page=1&idFilter=TAK-647-1001

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 20 investigative sites in the United States from 18 January 2023 to 30 December 2024.
Pre-assignment Details: A total of 11 participants were enrolled and received study treatment. The study was terminated early by the sponsor due to a strategic shift and reprioritization of clinical programs within Takeda.
Groups:
- Ontamalimab: Participants received ontamalimab 75 milligrams (mg) subcutaneous (SC) injection using a prefilled syringe once every 4 weeks (Q4W) on Day 1 and the last dose was administered at Week 20 with a total treatment period of 24 weeks.
Period: Overall Study
Arm/Group | Ontamalimab
Started | 11
Completed | 7
Not Completed | 4
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Population: The safety analysis set consisted of all participants who were enrolled in the study and had received at least 1 dose of study drug.
Groups:
- Ontamalimab: Participants received ontamalimab 75 mg SC injection using a prefilled syringe Q4W on Day 1 and the last dose was administered at Week 20 with a total treatment period of 24 weeks.
Arm/Group | Ontamalimab
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.3 (7.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An Adverse Event (AE) was defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. TEAEs was defined as any event that emerged or manifested at or after the initiation of treatment with a study drug or medicinal product, or any existing event that worsened in either intensity or frequency following exposure to the study drug or medicinal product.
Time Frame: From first dose of study drug up to Week 36
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Ontamalimab
Number analyzed (Participants) | 11
Participants | 6

2. Primary Outcome: Number of Participants With Clinically Significant Abnormalities in Clinical Laboratory Values
Description: Laboratory parameters included serum chemistry, hematology, urinalysis, and coagulation. Any Abnormality in clinical laboratory results which are deemed clinically significant by the investigator were reported.
Time Frame: From first dose of study drug up to Week 36
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Ontamalimab
Number analyzed (Participants) | 11
Participants
  Serum Chemistry | 0
  Hematology | 0
  Urinalysis | 0
  Coagulation | 0

3. Primary Outcome: Number of Participants With Clinically Significant Abnormalities in 12-lead Electrocardiogram (ECGs) Findings
Description: ECG included heart rate, QRS intervals, QT intervals, PR intervals, RR intervals and QT intervals corrected for heart rate using Fridericia's formula (QTcF) intervals parameters measurement. Any abnormality in ECG assessments which were deemed clinically significant by the investigator were reported.
Time Frame: From first dose of study drug up to Week 24
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Ontamalimab
Number analyzed (Participants) | 11
Participants | 0

4. Primary Outcome: Number of Participants With Clinically Significant Abnormalities in Vital Signs
Description: Vital signs included measurement of pulse rate, systolic, diastolic blood pressure, respiratory rate, Body mass index (BMI), body temperature and height. Any abnormality in vital signs which are deemed clinically significant by the investigator were reported.
Time Frame: From first dose of study drug up to 36 weeks
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Ontamalimab
Number analyzed (Participants) | 11
Participants | 0

5. Primary Outcome: Number of Participants With Clinically Significant Abnormalities in Body Weight
Description: Body weight was measured in kilograms (kg) at the specified time points. Any abnormality in body weight which are deemed clinically significant by the investigator were reported.
Time Frame: From first dose of study drug up to Week 36
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Ontamalimab
Number analyzed (Participants) | 11
Participants | 0

6. Secondary Outcome: Percent Change From Baseline in Pro-Collagen Type III (Pro-C3) Through Week 24
Description: Researchers measured the change in liver scarring using biomarkers. Biomarkers are substances measured in blood that show normal or abnormal activity taking place in the liver. Pro-C3 was measured in serum; Increasing levels indicate worsening of fibrosis activity. Blood samples were collected for assessment of Pro-C3 biomarker.
Time Frame: Baseline up to Week 24
Population: The full analysis set (FAS) consisted of all participants who were enrolled in the study, had received at least one dose of the study drug, and had at least one valid postbaseline assessment. Here, "Overall number of participants analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Ontamalimab
Number analyzed (Participants) | 8
percent change | -11.88 [-26.13 to 2.37]

7. Secondary Outcome: Percent Change From Baseline in Enhanced Liver Fibrosis (ELF) Through Week 24
Description: Researchers measured the change in liver scarring using biomarkers. Biomarkers are substances measured in blood that show normal or abnormal activity taking place in the liver. Blood samples were collected for an assessment of ELF score. The ELF score was calculated from the concentrations of the following serum biomarkers: tissue inhibitor of metalloproteinases- 1 (TIMP-1), procollagen III n-terminal propeptide (PIIINP), and hyaluronic acid (HA). ELF was a score on a scale of severity assessment against biopsy-proven fibrosis. A score of less than (<) 7.7 is none to mild, greater than (>) 7.7-9.8 is moderate, >9.8 is severe. Higher ELF scores represented worse disease outcome.
Time Frame: Baseline up to Week 24
Population: The FAS consisted of all participants who were enrolled in the study, had received at least one dose of the study drug, and had at least one valid postbaseline assessment. Here, "Overall number of participants analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Ontamalimab
Number analyzed (Participants) | 8
percent change | -0.13 [-3.61 to 3.35]

8. Secondary Outcome: Change From Baseline in Liver Iron-corrected T1 Mapping by Magnetic Resonance Imaging (cT1 MRI) at Week 24
Description: cT1 is a quantitative MRI relaxation parameter that measures liver inflammation and fibrosis. Participants underwent abdominal MRI to obtain liver cT1, which were used to assess fibro-inflammation. The change from baseline was calculated by subtracting the baseline values from the individual post-baseline values.
Time Frame: Baseline, Week 24
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: millisecond (ms)
Arm/Group | Ontamalimab
Number analyzed (Participants) | 10
millisecond (ms) | -32.0 (39.77)

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to Week 36
Arm/Group | Ontamalimab
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 6/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ontamalimab (N=11)
Abdominal pain upper (Gastrointestinal disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Dizziness (Nervous system disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Headache (Nervous system disorders) | 1
Hot flush (Vascular disorders) | 2
Hypertension (Vascular disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Tooth fracture (Injury, poisoning and procedural complications) | 1
Urinary tract infection (Infections and infestations) | 1
Vulvovaginal candidiasis (Infections and infestations) | 1

LIMITATIONS AND CAVEATS:
The study was terminated early by the sponsor due to a strategic shift and reprioritization of clinical programs within Takeda.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-09-18): https://cdn.clinicaltrials.gov/large-docs/82/NCT07052682/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-18): https://cdn.clinicaltrials.gov/large-docs/82/NCT07052682/SAP_001.pdf